CLINICAL TRIAL: NCT05733936
Title: Assessment of Biomechanical Determinants of Rehabilitation Protocols for ACL Reconstruction on the Quality of Performance and Risk of Reinjury: Randomized Controlled Trial
Brief Title: Biomechanical Determinants of Different Rehabilitation Protocols for ACL Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Omar Mohamed Ali Elabd, Lecturer of Orthopedics, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 004270
Record Dates: First submitted 2023-01-28; First posted 2023-02-17 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Knee Injuries; Rehabilitation
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- criterion-based rehabilitation protocol (Experimental): It's a three phases rehabilitation protocol with a goal-based progression which include a three criterion based postoperative phases: (1) impairment phase, (2) sport-specific training phase and (3) return to play phase. Patients can start with the next phase only if specific goals of the previous phase are achieved
  Interventions: Other: rehabilitation protocol
- accelerated rehabilitation protocol (Active Comparator): It's a four phases rehabilitation protocol mainly based on the remodeling process of the graft., emphasizing full passive knee extension, immediate weight bearing as tolerated and functional exercises
  Interventions: Other: rehabilitation protocol

INTERVENTIONS:
Other: rehabilitation protocol — rehabilitation protocols after ACLR have been described, aiming to improve muscle strength and knee stability through muscle strengthening exercises in addition to exercises to improve joint proprioception

SUMMARY:
Purpose of the study is to investigate the effects of the criterion rehabilitation protocol versus accelerated rehabilitation protocol on the biomechanical determinants of the quality of performance and risk of reinjury.

ELIGIBILITY:
Inclusion Criteria:

* Amateur male athletes who underwent ACLR surgery with an autologous hamstring (HS) graft.
* Ranging in age from 18 to 35 years.
* Underwent a pre-operative rehabilitation program with minimal knee effusion, full Extension, good patellofemoral mobility
* Ability to actively control the quadriceps.

Exclusion Criteria:

* ACLR with any graft other than a hamstring graft
* ACL revision surgery
* associated medial or lateral ligamentous injuries
* previous meniscectomy or meniscal repair
* simultaneous meniscectomy or meniscus repair with the ACLR
* cartilage damage.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dynamic knee valgus during Single leg landing-jump test using CLINICAL CLIMA 3DMA | 15 minutes
  From the coronal plane, dynamic knee valgus is the angle of the knee
Lateral trunk flexion during Single leg landing-jump test using CLINICAL CLIMA 3DMA | 15 minutes
  From the coronal plane, trunk lateral flexion angle is the angle of the trunk
knee flexion angle during Single leg landing-jump test using CLINICAL CLIMA 3DMA | 15 minutes
  From sagittal plane, knee flexion angle is the angle of the knee

CONTACTS AND LOCATIONS:
Locations (1):
- Delta university, Gamasa, Eldakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: No